CLINICAL TRIAL: NCT01495741
Title: An Observational Post-Authorization Safety Surveillance (PASS) Study of Sycrest® (Asenapine) Among Patients Aged 18 and Older Diagnosed With Bipolar Disorder
Brief Title: Post-Authorization Safety Surveillance Study of Asenapine in Participants With Bipolar Disorder (P08307)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P08307; MK-8274-110 (Other: Merck)
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Mania; Manic; Depressive; Manic Depressive
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Mania

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asenapine: Participants prescribed asenapine
- Risperidone Comparator: Participants prescribed risperidone
- Olanzapine Comparator: Participants prescribed olanzapine

SUMMARY:
This study will assess asenapine (Sycrest®) use in participants with bipolar disorder; comparison will be made to the use of risperidone (RISPERDAL®CONSTA®) and olanzapine (Zyprexa®). The occurrence of identified and potential clinically important risks will also be assessed.

ELIGIBILITY:
Inclusion Criteria for the Bipolar Disease Cohort:

* A diagnosis of Bipolar Disorder

Exclusion Criteria for the Bipolar Disease Cohort:

* None

Inclusion Criteria for the potential Schizophrenia Cohort:

* A diagnosis of schizophrenia

Exclusion Criteria for the potential Schizophrenia Cohort:

* A prior and/or concomitant diagnosis of bipolar disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Bipolar Disorder codes who are included in the United Kingdom Clinical Practice Research Datalink (CPRD) and, if required, The Health Improvement Network (THIN) database.
  If pre-specified sample size and exposure criteria are met, secondary objectives will be conducted in 2 separate study populations: 1. Participants treated with asenapine and diagnosed with schizophrenia and no prior and/or concomitant diagnosis of bipolar disorder; 2. Participants treated with asenapine with no prior and/or concomitant diagnoses of bipolar disorder or schizophrenia, but diagnosed with i) Alzheimer's disease, ii) other diagnoses - mental disorders or iii) no diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Bipolar Disorder with Identified and Potential Clinically Important Risks | Approximately 1 year
  Identified and potential clinically important risks will include: extrapyramidal symptoms, somnolence and sedation, neuroleptic malignant syndrome, rhabdomyolysis, seizure, hyperprolactinaemia, orthostatic hypotension, neutropenia, allergic reactions, dyslipidaemia and diabetes mellitus with the use of asenapine versus risperidone or olanzapine

SECONDARY OUTCOMES:
Number of Participants with Schizophrenia with Identified and Potential Clinically Important Risks | Approximately 1 year
  When enrollment and participant exposure reaches a level that adequate power (80%) is achieved according to pre-defined power calculations, risk incidence with use of asenapine in participants diagnosed with schizophrenia with no prior and/or concomitant diagnosis of bipolar disorder will be analyzed. Identified and potential clinically important risks will include: extrapyramidal symptoms, somnolence and sedation, neuroleptic malignant syndrome, rhabdomyolysis, seizure, hyperprolactinaemia,orthostatic hypotension, neutropenia, allergic reactions, dyslipidaemia and diabetes mellitus with the use of asenapine versus risperidone or olanzapine
Number of Participants without Diagnoses of Schizophrenia or Bipolar Disorder with Identified and Potential Clinically Important Risks | Approximately 1 year
  When enrollment and participant exposure reaches a level that adequate power (80%) is achieved according to pre-defined power calculations, risk incidence with use of asenapine in participants with no prior and/or concomitant diagnoses of bipolar disorder or schizophrenia, but diagnosed with i) Alzheimer's disease, ii) other diagnoses - mental disorders or iii) no diagnosis, will be analyzed. Identified and potential clinically important risks will include: extrapyramidal symptoms, somnolence and sedation, neuroleptic malignant syndrome, rhabdomyolysis, seizure, hyperprolactinaemia,orthostatic hypotension, neutropenia, allergic reactions, dyslipidaemia and diabetes mellitus with the use of asenapine

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC